CLINICAL TRIAL: NCT05742789
Title: Effect of Anesthetics on Troponin I and С-reactive Protein in Mitral, Tricuspid and Aortic Valve Replacement/Plastic in Adult: a Randomized Clinical Study
Brief Title: Effect of Anesthetics on Troponin I and С-reactive Protein
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astana Medical University (Other)
Responsible Party: Principal Investigator, Bekzat Baiterek, Clinical Professor, Astana Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 6
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Mitral Valve Insufficiency; Aortic Valve Insufficiency; Cardiac Disease
Keywords: Mitral Valve Insufficiency; Aortic Valve Insufficiency; Troponin I; propofol; isoflurane; sevoflurane
MeSH Terms: conditions — Mitral Valve Insufficiency; Aortic Valve Insufficiency; Heart Diseases | interventions — Propofol; Isoflurane; Sevoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Propofol (Other): Anesthesia
  Interventions: Drug: Propofol
- Isofluran (Other): Anesthesia
  Interventions: Drug: Isoflurane
- Sevofluran (Other): Anesthesia
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — To maintain anaesthesia in Group 1 P, propofol was used as an anaesthetic in a dose of 4-6 mg/kg/h intravenously on a perfusor
  Other Names: Propofol;
  Arms: Propofol
Drug: Isoflurane — В качестве анестетика использовали изофлуран - 1,1-1,2 MAC.
  Arms: Isofluran
Drug: Sevoflurane — в качестве анестетика использовали севофлуран в дозе - 1,7-1,9 ПДК.
  Arms: Sevofluran

SUMMARY:
Abstract Troponin is one of the cardiac biomarkers and its high level correlates to high risk of cardiac myocytes damage. C-reactive protein (CRP) in cardiosurgery participates in the Systemic Inflammation Response Syndrome, and heart-lung apparatus is a powerful stimulator of the systemic inflammatory reaction.

Objective: To assess effect of anesthetics on troponin I and СRP in mitral, tricuspid and aortic valve replacement/plastic in adult.

Methods. Single-center prospective randomized controlled clinical study. A total of 95 patients were assigned randomly into three groups according to the type of anesthesia: the first group of 32 patients with propofol, the second group with sevoflurane - 32 patients, and the last - 31 patients were with isoflurane.

Levels of the cardiac troponin I were calculated in ng/ml с using a portable fluorometric analyzer I-CHROMAII, manufacture of BoditechMedInc (South Korea). Normal range: <0.04 ng/ml. CRP concentration in plasma has been determined using a biochemical analyzer Biosystems BA-200 (Spanish company, Barcelona) according to the manufacturer's instructions. The normal level of CRP is less than 5 mg/l.

DETAILED DESCRIPTION:
The examination and treatment data of 95 patients operated in the departments of cardiovascular surgery of the City multidisciplinary hospital No. 2 were included in the study. All patients underwent mitral, aortic, tricuspid valve replacement/plasty under cardiopulmonary bypass (CPB) conditions. This research work was conducted between 2021 and 2023. To calculate the sample size, we used the formula n=t2*D*N/confidence interval*N+t2*α, which will allow to identify the static significance of the study.

Inclusion criteria: insufficiency of mitral, tricuspid and aortic valves of 3-4th degree; only planned surgeries; age range 40-60 years old; patients corresponding to II-III grade according to the scale of the American Society of Anaesthesiologists.

Exclusion criteria: pregnancy; acute coronary syndrome; hemodynamic instability.

All patients were assigned randomly into three groups according to the type of anesthesia: the first group of 32 patients with propofol, the second group with sevoflurane - 32 patients, and the last - 31 patients were with isoflurane.

The level of cardiac troponin I were calculated in ng/ml using a portable fluorometric analyzer i-CHROMAII, production of BoditechMedInc (South Korea). The normal range: <0.04 ng/ml. The analyzer Triage® Meter Pro of Alere San Diego Inc. production (USA).

Three blood samples were taken in the patients before the anaesthesia, in 12 hours post-surgery and in 48 hours post-surgery. Blood samples were taken in the sterile test-tubes, containing no EDTA and heparin, centrifugated and stored at temperature -20 °С to avoid the erroneously low results.

CRP concentrations in plasma were determined using the biochemical analyzer Biosystems BA-200 (Spanish company, Barcelona) according to the manufacturer's instructions. The normal level of CRP is less than 5 mg/l. Blood samples were taken in the patients before the anaesthesia, 1st day post-surgery, 3rd and 5th days post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* The age is between 50-65 years old;
* Mitral and aortic valve insufficiency grade 3-4;
* Participants of both sexes will be included in the study;
* Planned surgical interventions;
* Signed informed consent.

Exclusion Criteria:

* pregnancy (risk to the baby and mother)
* hypertensive disease
* coronary artery disease;
* current unstable angina pectoris;
* preoperative hemodynamic instability, defined as the use of vasopressors;

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Troponin I | 2 year
  Cardiac troponin I levels were calculated in ng/mL using the i-CHROMAII portable fluorescent analyzer manufactured by BoditechMedInc. (South Korea). Normal range: <0.4 ng/mL.
С-reactive protein | 2 year
  С-reactive protein concentrations in plasma were determined using the biochemical analyzer Biosystems BA-200 (Spanish company, Barcelona) according to the manufacturer's instructions.

CONTACTS AND LOCATIONS:
Overall Officials: Alibek Kh Mustafin, Professor, Study Director — Astana Medical University
Locations (1):
- Bekzat, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: No